CLINICAL TRIAL: NCT06118996
Title: Comparing the Efficacy of 3D Ultrasound Imaging of Breast Pathology Between a Custom ITA Device and Invenia™ ABUS System by GE Medical
Brief Title: Breast 3DUS ABUS System Comparison
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14144
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Diseases
Keywords: 3D Ultrasound; Intervention
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients at Risk of Breast Cancer (Experimental): These patients will be imagined with an experimental device designed to acquire ultrasound in three dimensional volumes
  Interventions: Device: 3D Ultrasound Image Acquisition

INTERVENTIONS:
Device: 3D Ultrasound Image Acquisition — A custom device will be used with a clinical ultrasound machine to acquire ultrasound images of the breast.

SUMMARY:
This comparative study will recruit 30 females who are scheduled for mammography and ultrasound assessment. The clinical 2D ultrasound is performed routinely, and the research portion of this study will add a few extra 3-D ultrasound images during the procedure. The ultrasound imaging laboratory under the direction of Dr. Aaron Fenster has developed a customized device designed to acquire 3D ultrasound of the breast using a commercial ultrasound machine. The purpose is to see how well 3-dimensional ultrasound acquire from that device is able to visualize tumours and other key features in comparison to the clinical system InveniaTM developed by GE Medical.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients who are scheduled for screening ABUS
* Adults Patients who are scheduled for short term follow-up with ABUS.
* Must be at least 18 years of age or older.
* Must be proficient in English (reading/writing).

Exclusion Criteria:

* Patients with breast implants.
* Patients with contraindication for ABUS.
* Patients who cannot tolerate ABUS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Breast Images | 24 months
  Images of the breast anatomy will be compared to standard of care imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No